CLINICAL TRIAL: NCT01403038
Title: A Phase 1, Open-Label Study of the Effects of Elagolix on Ovarian Activity, Ovulation and Ovarian Reserve in Premenopausal Females
Brief Title: An Open-label Study of the Effects of Elagolix in Adult Premenopausal Females
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: AbbVie (prior sponsor, Abbott) (Industry)
Collaborators: Neurocrine Biosciences (Industry)
Responsible Party: Sponsor
Organization: AbbVie (Industry)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Basic Science
Other Study IDs: M12-673
Record Dates: First submitted 2011-06-01; First posted 2011-07-27 (Estimated); Last update posted 2013-01-08 (Estimated); Status verified 2013-01

CONDITIONS: Folliculogenesis
Keywords: healthy volunteers; elagolix; endometriosis; ovarian reserve; gonadotropin-releasing hormone antagonist; ovulation; ovarian activity
MeSH Terms: conditions — Endometriosis | interventions — elagolix

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (7):
- Elagolix Dose Regimen 1 (Experimental): Elagolix Dose regimen 1 for 84 days
  Interventions: Drug: Elagolix
- Elagolix Dose Regimen 2 (Experimental): Elagolix Dose Regimen 2 for 84 days
  Interventions: Drug: Elagolix
- Elagolix Dose Regimen 3 (Experimental): Elagolix Dose Regimen 3 for 84 days
  Interventions: Drug: Elagolix
- Elagolix Dose Regimen 4 (Experimental): Elagolix Dose Regimen 4 for 84 days
  Additional Dose Regimens may be added and will be administered for 84 days.
  Interventions: Drug: Elagolix
- Elagolix Dose Regimen 5 (Experimental): Elagolix Dose Regimen 5 for 84 days
  Interventions: Drug: Elagolix
- Elagolix Dose Regimen 6 (Experimental): Elagolix Dose Regimen 6 for 84 days
  Interventions: Drug: Elagolix
- Elagolix Dose Regimen 7 (Experimental): Elagolix Dose Regimen 7 for 84 days
  Interventions: Drug: elagolix

INTERVENTIONS:
Drug: Elagolix — Elagolix Dose Regimen 1 for 84 days
  Other Names: ABT-620, elagolix sodium
  Arms: Elagolix Dose Regimen 1
Drug: Elagolix — Elagolix Dose Regimen 2 for 84 days
  Other Names: ABT-620, elagolix sodium
  Arms: Elagolix Dose Regimen 2
Drug: Elagolix — Elagolix Dose Regimen 3 for 84 days
  Other Names: ABT-620, elagolix sodium
  Arms: Elagolix Dose Regimen 3
Drug: Elagolix — Elagolix Dose Regimen 4 for 84 days Other interventions may be added
  Other Names: ABT-620, elagolix sodium
  Arms: Elagolix Dose Regimen 4
Drug: Elagolix — Elagolix Dose Regimen 5 for 84 days
  Other Names: ABT-620, elagolix sodium
  Arms: Elagolix Dose Regimen 5
Drug: Elagolix — Elagolix Dose Regimen 6 for 84 days
  Other Names: ABT-620, elagolix sodium
  Arms: Elagolix Dose Regimen 6
Drug: elagolix — Elagolix plus Activella Dose Regimen 7 for 84 days
  Other Names: ABT-620, elagolix sodium
  Arms: Elagolix Dose Regimen 7

SUMMARY:
This is an open-label Phase 1 study in healthy premenopausal females evaluating the effects of different dosing regimens of elagolix on ovarian activity, ovulation, and ovarian reserve and to assess the effect of elagolix on selected endocrine/hormone levels.

DETAILED DESCRIPTION:
This is an open-label, multiple-dose, Phase 1 study in premenopausal subjects aged 18 years to 40 years, with a history of regular menstrual cycles (24 to 32 days long) and no evidence of significant gynecological disorders. The objective of the study is to determine the effects of different dosing regimens of elagolix on ovulation, ovarian activity, and ovarian reserve. The study consists of 3 periods: a Screening Period of up to 50 days prior to the first dose, a Treatment Period of 3 months duration (Cycles 1-3), and a Follow-up Period of up to 60 days. During the Screening and Treatment menstrual cycles, serial transvaginal ultrasounds and determination of serum levels of luteinizing hormone, follicle-stimulating hormone, estradiol, progesterone, and inhibin B will be performed three times weekly. Subjects will maintain a daily diary of uterine bleeding. Pregnancy testing will be performed frequently throughout the study. Subjects will be required to use nonhormonal dual contraception consistently during the study, and will be counseled on appropriate and effective forms of birth control to promote pregnancy prevention.

ELIGIBILITY:
Inclusion Criteria:

- Premenopausal female, between 18 and 40 years of age, inclusive - History of regular menstrual cycles - Endocrine and ultrasonographic evidence of ovulation and normal ovulatory cycle during the screening period - Follicle-stimulating hormone level of <35 mIU/mL - Agrees to use required birth control methods during the entire length of participation in the study

Exclusion Criteria:

- Screening ultrasound results show a clinically significant gynecological disorder - Surgical history of hysterectomy without oophorectomy, unilateral or bilateral oophorectomy, removal of ovarian cysts - Less than 6 months postpartum or post-lactation at the start of study drug dosing - Pregnant or breast feeding or is planning a pregnancy within the next 12 months - Testosterone concentration >120 ng/dL at screening

Ages: 18 Years to 40 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 216 (Actual)
Dates: Start 2011-06; Primary Completion 2012-10 (Actual); Study Completion 2012-11 (Actual)

PRIMARY OUTCOMES:
Ovulation Classification | During the baseline menstrual cycle and monthly during the treatment cycles 1, 2, and 3 for up to month 3.
  Presence or absence of ovulation
Ovarian Activity | During the baseline menstrual cycle and monthly during the treatment cycles 1, 2, and 3 for up to month 3.
  As measured by the Hoogland and Skouby 6-point ovarian activity grading system

SECONDARY OUTCOMES:
Endocrine Parameters | During the 16 week study period (4 week screening period and 12 week treatment period) for up to month 3
  Estuarial, Progesterone, luteinizing hormone, follicle stimulating hormone
Ovarian Reserve | During the baseline menstrual cycle and monthly during the treatment cycles 1, 2, and 3 for up to month 3.
  Inhibin-B and Antimullerian hormone
Adverse events | All adverse events occurring through the Final Visit will be reported
  All adverse events will be collected by subject self-report and review of laboratory parameters, physical exam. vital sign measurements and electrocardiograms.
Clinical Laboratory Tests | Change from baseline to Cycles 1, 2, and 3 or Final Visit
  Chemistry, hematology, urinalysis
12-lead Electrocardiogram | Change from baseline to Week 4 and Final Visit
  12-lead Electrocardiogram
Vital Signs | Change from baseline to Cycles 1, 2, and 3 or Final Visit
  Blood pressure, heart rate, temperature

CONTACTS AND LOCATIONS:
Overall Officials: Kristof Chwalisz, MD, PhD, MD, Study Director — AbbVie
Locations (22):
- United States (20):
  - Site Reference ID/Investigator# 50805, Colorado Springs, Colorado
  - Site Reference ID/Investigator# 51270, Colorado Springs, Colorado
  - Site Reference ID/Investigator# 50884, Denver, Colorado
  - Site Reference ID/Investigator# 50404, Lonetree, Colorado
  - Site Reference ID/Investigator# 50904, Miami, Florida
  - Site Reference ID/Investigator# 50402, South Miami, Florida
  - Site Reference ID/Investigator# 50808, Tampa, Florida
  - Site Reference ID/Investigator# 50807, Naperville, Illinois
  - Site Reference ID/Investigator# 50804, Oak Brook, Illinois
  - Site Reference ID/Investigator# 50762, Durham, North Carolina
  - Site Reference ID/Investigator# 50403, Winston-Salem, North Carolina
  - Site Reference ID/Investigator# 50810, Cincinnati, Ohio
  - Site Reference ID/Investigator# 50883, Portland, Oregon
  - Site Reference ID/Investigator# 50803, Philadelphia, Pennsylvania
  - Site Reference ID/Investigator# 51546, Philadelphia, Pennsylvania
  - Site Reference ID/Investigator# 50806, San Antonio, Texas
  - Site Reference ID/Investigator# 51342, San Antonio, Texas
  - Site Reference ID/Investigator# 50811, Sandy City, Utah
  - Site Reference ID/Investigator# 50902, Norfolk, Virginia
  - Site Reference ID/Investigator# 50882, Seattle, Washington
- Puerto Rico (2):
  - Site Reference ID/Investigator# 53363, San Juan
  - Site Reference ID/Investigator# 53362, Santurce

REFERENCES:
- [Derived] Archer DF, Ng J, Chwalisz K, Chiu YL, Feinberg EC, Miller CE, Feldman RA, Klein CE. Elagolix Suppresses Ovulation in a Dose-Dependent Manner: Results From a 3-Month, Randomized Study in Ovulatory Women. J Clin Endocrinol Metab. 2020 Mar 1;105(3):dgz086. doi: 10.1210/clinem/dgz086. PMID 31650182
- [Derived] Winzenborg I, Nader A, Polepally AR, Liu M, Degner J, Klein CE, Mostafa NM, Noertersheuser P, Ng J. Population Pharmacokinetics of Elagolix in Healthy Women and Women with Endometriosis. Clin Pharmacokinet. 2018 Oct;57(10):1295-1306. doi: 10.1007/s40262-018-0629-6. PMID 29476499